CLINICAL TRIAL: NCT05910008
Title: Evaluation of Intraoperative O-ARM Stereotactic Imaging Versus Conventional Pre-operative Stereotactic Imaging in Deep Brain Stimulation for Parkinson's Disease
Brief Title: O-ARM Stereotactic Imaging in Deep Brain Stimulation for Parkinson's Disease
Acronym: STEREOBLOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/22/0489; 2023-A00871-44 (Other: ID-RCB)
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: Stereotactic imaging; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- O-Arm stereotactic imaging (Experimental): Imaging is performing directly in the operating room.
  Interventions: Procedure: O-Arm Stereotactic imaging
- Standard stereotactic imaging (Active Comparator): Imaging is performing in Radiology department.
  Interventions: Procedure: Standard Stereotactic imaging

INTERVENTIONS:
Procedure: O-Arm Stereotactic imaging — Prior to electrode implantation, O-ARm stereotactic imaging (Magnetic Resonance Imaging)
  Arms: O-Arm stereotactic imaging
Procedure: Standard Stereotactic imaging — Prior to electrode implantation, standard stereotactic imaging (Magnetic Resonance Imaging)
  Arms: Standard stereotactic imaging

SUMMARY:
During deep brain stimulation procedures in Parkinson's disease (PD), the most important prognostic element is the positioning of the surgical electrode in the subthalamic nucleus which is the anatomical target. The main objective of this project is therefore to compare 2 techniques thanks to a prospective comparative randomised open-label study: the use of O-ARM to acquire stereotactic imaging directly in the operating room and the standard technique requiring stereotactic imaging to be performed in the radiology department.

DETAILED DESCRIPTION:
Prior to electrode implantation we perform stereotactic imaging which requires the fixation of a stereotactic frame on the patient's head before imaging (Magnetic Resonance Imaging MRI / Computed Tomography CT). Currently, it is necessary to transfer the patient to the imaging department outside of the operating room after the stereotactic frame has been placed, for imaging (either MRI or CT) and then to return to the operating room to begin the electrode implantation procedure. Since 2016, the new generation O-Arm 2 allows the acquisition of stereotactic imaging with the stereotactic frame in place by increasing the field of view (40 cm versus 20 cm previously) directly in the operating room. As a result, the transfer step to the MRI and CT scanner preoperatively may no longer be necessary, and the procedure can be started more quickly with greater comfort and safety for the patient and the anaesthesia team. Several teams around the world have begun to use framed O-Arm as the gold standard for stereotactic imaging. However, no randomised controlled study has been performed to date comparing O-Arm stereotactic imaging with pre-operative CT and/or MRI reference imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of idiopathic Parkinson's disease at the stage of motor fluctuations despite optimal medical treatment
* Indication for Deep Brain Stimulation (DBS) of the subthalamic nucleus approved by the local multidisciplinary deep brain stimulation committee after an operability assessment (see Appendix)
* Informed and signed patient consent
* Affiliation to a social security scheme

Exclusion Criteria:

* Significant cognitive decline assessed in a dedicated multidisciplinary consultation
* Contraindication to Magnetic Resonance Imaging (MRI)
* Presence of pathologies contraindicating deep brain stimulation
* No contraceptive treatment for women of childbearing age
* Pregnant or breastfeeding woman
* Anticoagulant or antiaggregant treatment that cannot be stopped
* Persons under legal protection (persons deprived of liberty or incapable of giving consent or under guardianship or tutelage...)
* Patient with severe psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
The absolute accuracy of Deep Brain Stimulation electrode implantation | 48 hours
  The radial distance between the theoretical target and the electrode in the plane of the target regardless of the chosen trajectory (central, anterior, lateral). This distance corresponds to the minimum error between the target and the electrode. This measurement is made from the postoperative brain scan.

SECONDARY OUTCOMES:
The anatomical accuracy of Deep Brain Stimulation electrode implantation | 48 hours
  Automatic calculation of the vector distance between the middle of pad 1 on the electrode and the theoretical target by software.
Central and alternate position of the electrodes rate | 1 day
  Comparison of the anatomical location of the electrode compared to the anatomical target (subthalamic nucleus) after matching preoperative Magnetic Resonance Imaging (MRI) images
Surgical Times | 1 day
  Time from the end of the stereotactic frame to the surgical incision and time from the entry into room to the exit from room after generator implantation.
Clinical effectiveness | 6 months
  Comparison of The Unified Parkinson's Disease Rating Scale (UPDRS) II, III and IV scores between baseline and 6 months and then at 6 months between the 2 groups.
  The UPDRS scale is composed of 47 items grouped into three parts : II, III and IV. Responses scale ranging from 0 (normal/no symptoms) to 4 (severe).
Daily dose of Levodopa decrease | 6 months
  The change in Levodopa Equivalent Daily Dose (LEDD) before surgery and at 6 months compared between the 2 groups. This LEDD corresponds to the amount of antiparkinsonian treatments prescribed to the patient
Adverse effect rate | 6 months
  Clinical reporting of patient events/adverse reactions
Correlation between absolute accuracy and clinical effectiveness | 6 months
  Correlation between radial accuracy and UPDRS score for both groups

CONTACTS AND LOCATIONS:
Overall Officials: Amaury De Barros, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France